CLINICAL TRIAL: NCT03413033
Title: Immediate Effects of Two Semi-occluded Vocal Tract Exercises on Laryngeal Activity of Individuals With Constant Vocal Effort
Brief Title: Immediate Effects of Two Semi-occluded Vocal Tract Exercises
Status: Completed | Type: Observational
Sponsor: Universidad Nacional de Colombia (Other)
Responsible Party: Principal Investigator, Andres Fernando Delprado, Msc Physiology Student, Universidad Nacional de Colombia
Other Study IDs: 012-210-18
Record Dates: First submitted 2018-01-18; First posted 2018-01-29 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: Voice
Keywords: Semi-occluded vocal tract; resonance tubes; tongue trill; voice therapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: 43 participants will produce the vowel /a:/ three times as baseline during 5 seconds in habitual, comfortable speaking pitch and loudness. Thereafter, participants will produce series of a semi-occluded vocal tract exercises (resonance tube or lip trill). Afterwards, subjects will produce the vowel /a:/ three times once again. Electroglottographic signals will be captured before and after each exercise. A 15 minutes voice rest will be taken between exercises by all subjects.
  Interventions: Other: Resonance tube; Other: Tongue trill

INTERVENTIONS:
Other: Resonance tube — Participants will phonate into a tube (10cm length 4mm inner diameter) during 5 minutes. They will produce series of the vowel /u/ into the tube. They will be asked to maintain the same pitch and loudness as they did in the baseline samples. They will be perceptually controlled by experimenters. When performing the exercise, the participants will be instructed to phonate with ease voice and to sense vibrations in the anterior face and the mouth.
Other: Tongue trill — Participants will produce series of a similar /r/ Spanish sound during 5 minutes. They will be asked to maintain the same pitch and loudness as they did in the baseline samples. They will be perceptually controlled by experimenters. When performing the exercise, the participants will be instructed to phonate with ease voice and to sense vibrations in the anterior face and the mouth.

SUMMARY:
This study aims to observe the physiological effects of two different Semi-occluded vocal tract (SOVT) exercises in the larynx when they are executed by individuals with constant vocal effort and without vocal pathology.

DETAILED DESCRIPTION:
SOVT is a voice education or rehabilitation method that involves different postures which partially occlude or elongate the vocal tract. It causes a change in the vibration pattern of the vocal folds. SOVT postures have been postulated to produce changes in contact quotient (CQ), measured with electroglottograph (EGG). This study aims to observe the physiological effects of two different SOVT exercises in larynx when they are executed by people with constant vocal effort and without vocal pathology. In order to do so, EGG will be performed before and after 43 volunteers execute two SOVT exercises (tongue trill and resonance tubes). The following parameter will be captured: CQ. A t-paired test will be performed to compare pre and post-test information. Furthermore, a generalized estimating equation will be fit to find the effects of each exercise in the subjects.

This protocol was modified due to different administrative issues related to the use of the stroboscopy (one of the assesment tools previosly considered), so that stroboscopy was removed from the protocol.

ELIGIBILITY:
Inclusion Criteria:

* No current or past history of voice disorders.
* No current or past voice training or therapy.
* Vocal use larger than 20 hours per week.

Exclusion Criteria:

* Laryngeal pathology during execution of stroboscopy.
* Flu-like symptoms during measures.
* Trouble with execution of semi-occluded vocal tract exercises.
* Allergy to electrodes.

Ages: 25 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy university teachers despite constant vocal effort, without past voice training or therapy.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2018-08-16 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Contact quotient (CQ) | 1 hour
  Improvement of vocal folds vibration pattern, demonstrated by a decrease of the mean CQ, measured with Electroglottography.

CONTACTS AND LOCATIONS:
Overall Officials: Luisa F Ángel Gordillo, Study Director — Universidad Nacional de Colombia
Locations (1):
- Universidad Nacional de Colombia, Bogotá, Colombia

IPD SHARING:
Plan to Share IPD: No